CLINICAL TRIAL: NCT04032938
Title: Clinical and Multi-omics Study on Gut Microbiota in Critical Ill Patients After Cardiovascular Surgery Combined Cardiopulmonary Bypass With or Without Sepsis（CPB-MUL-GM Study): a Prospective Study Protocol
Brief Title: Multi-omics Study on Gut Microbiota in Critical Ill Patients After Cardiopulmonary Bypass
Acronym: CPB-MUL-GM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wenyan Ding, Department of Critical Care Medicine，Doctor in Reading, Peking Union Medical College Hospital
Other Study IDs: ZS-1612
Record Dates: First submitted 2019-07-07; First posted 2019-07-25 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Sepsis; Cardiopulmonary Bypass
Keywords: Cardiopulmonary Bypass; Gastrointestinal Microbiome; Thoracic Surgery; Metagenomics; Metabolomics; sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Feces and blood samples will be obtained and stored at -80℃.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the control group: 30 healthy people as the control group.
- the case group: 60 patients were admitted to intensive care unit (ICU) as the case group after cardiac surgery and extracorporeal circulation. This group should contain 30 patients with fever and/or hemodynamic instability and 30 patients with normothermia and normal hemodynamic.
  Interventions: Procedure: extracorporeal circulation during cardiac surgery

INTERVENTIONS:
Procedure: extracorporeal circulation during cardiac surgery — We will observe the cardiopulmonary bypass status and time of patients undergoing cardiac surgery and extracorporeal circulation due to their medical needs.
  Groups: the case group

SUMMARY:
Using metagenomics as well as metabolomics, the variation of the gut microbiota and host metabolite profiles of patient after undergoing CPB were explored.

DETAILED DESCRIPTION:
This protocol is designed as a prospective observational case-control study in patients who underwent cardiopulmonary bypass (CPB) due to cardiac surgery. 30 healthy persons were selected as control group. The case group included patients admitted to intensive care unit (ICU) after cardiac surgery and extracorporeal circulation which is performed by the Department of cardiac surgery of Peking Union Medical College Hospital. The patients enrolled should be divided into two groups according to their primary outcomes: one grouped fever and/or hemodynamic instability after cardiopulmonary bypass and the other grouped normothermia and normal hemodynamic during 48 hours after surgery(cause an infection manifested >48 hours after admission was defined as hospital acquired. ). Sample collection was terminated when both groups received 30 cases. These 60 cases would regard as the case group. Additionally, all the CPB patients we observed will be divided into survivors and non-survivors based on the 28-day survival. Feces and blood samples will be obtained at certain time points（initial sampling at least one day before the surgery, repeat sampling within 24-48 hours after CPB）. The fecal samples analysis will apply metagenomics and the feces and blood samples will be analyzed using untargeted metabolomics method. In this study, the stratification of gut microbial communities in patients underwent extracorporeal circulation were explored and analysed the variation of metabolite in patients's plasma and fecal samples. Predictive bio-markers and possible pathogenesis of fever and/or hemodynamic instability after CPB will be also provided by clinical outcomes analysis combined with multi-omics study.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be admitted to ICU between 18 and 85 years of age who will undergo extracorporeal circulation during cardiac surgery and provided written informed consent will be enrolled as candidates of case group.
* Healthy volunteers will be enrolled as control group.

Exclusion Criteria:

* Patients had a fever before surgery, regardless of the etiological evidence of infection;
* had anti-infective treatment before surgery;
* had gastrointestinal surgery which left the digestive system dysfunctional;
* had a history of CPB in 6 month;
* reject or abandon ICU therapeutic intervention.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 healthy volunteers will be randomly selected as the control group.
  Patients enrolled in the case group underwent cardiac surgery combined with extracorporeal circulation for medical reasons.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Surgery | During sample collection
  cardiovascular surgery with cardiopulmonary bypass VS. non-surgery non-surgery is defined as healthy people who don't need surgery.

SECONDARY OUTCOMES:
Anal temperature | within 24-48 hours after cardiopulmonary bypass
  Fever VS. non-fever
  Definition:
  Fever: The axillary body temperature is over 38.3℃. Non-fever: The axillary body temperature is below or equal to 38.3℃.
Hemodynamics | within 24-48 hours after cardiopulmonary bypass
  Hemodynamic instability VS. normal hemodynamic
  Definition:
  Hemodynamic instability: Vasopressor therapy needed to elevate MAP (mean artarial pressure) ≥65 mmHg.
survival | within 28 days after CPB
  survivors vs. non-survivors survivor: Patients survive for 28 days or more after CPB. non-survivors: Patients survive less than 28 days after CPB.

CONTACTS AND LOCATIONS:
Overall Officials: Longxiang Su, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Peking Union Medical College and Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
After the trial is completed, we may publish the IPD in the paper.

REFERENCES:
- [Background] Sergeant P, de Worm E, Meyns B. Single centre, single domain validation of the EuroSCORE on a consecutive sample of primary and repeat CABG. Eur J Cardiothorac Surg. 2001 Dec;20(6):1176-82. doi: 10.1016/s1010-7940(01)01013-2. PMID 11717024
- [Background] Ariyaratnam P, Ananthasayanam A, Moore J, Vijayan A, Hong V, Loubani M. Prediction of Postoperative Outcomes and Long-Term Survival in Cardiac Surgical Patients Using the Intensive Care National Audit & Research Centre Score. J Cardiothorac Vasc Anesth. 2019 Nov;33(11):3022-3027. doi: 10.1053/j.jvca.2019.05.034. Epub 2019 May 27. PMID 31227375
- [Background] Gorski A, Hamouda K, Ozkur M, Leistner M, Sommer SP, Leyh R, Schimmer C. Cardiac surgery antibiotic prophylaxis and calculated empiric antibiotic therapy. Asian Cardiovasc Thorac Ann. 2015 Mar;23(3):282-8. doi: 10.1177/0218492314546028. Epub 2014 Jul 24. PMID 25061221
- [Background] Wang YC, Wu HY, Luo CY, Lin TW. Cardiopulmonary Bypass Time Predicts Early Postoperative Enterobacteriaceae Bloodstream Infection. Ann Thorac Surg. 2019 May;107(5):1333-1341. doi: 10.1016/j.athoracsur.2018.11.020. Epub 2018 Dec 12. PMID 30552885
- [Background] A. F. Ueber peritoneale infection. Wien Klin Wochenschr. 1891;4:241, 265, 285.
- [Background] Dickson RP, Singer BH, Newstead MW, Falkowski NR, Erb-Downward JR, Standiford TJ, Huffnagle GB. Enrichment of the lung microbiome with gut bacteria in sepsis and the acute respiratory distress syndrome. Nat Microbiol. 2016 Jul 18;1(10):16113. doi: 10.1038/nmicrobiol.2016.113. PMID 27670109
- [Background] Singer BH, Dickson RP, Denstaedt SJ, Newstead MW, Kim K, Falkowski NR, Erb-Downward JR, Schmidt TM, Huffnagle GB, Standiford TJ. Bacterial Dissemination to the Brain in Sepsis. Am J Respir Crit Care Med. 2018 Mar 15;197(6):747-756. doi: 10.1164/rccm.201708-1559OC. PMID 29232157
- [Background] Ojima M, Motooka D, Shimizu K, Gotoh K, Shintani A, Yoshiya K, Nakamura S, Ogura H, Iida T, Shimazu T. Metagenomic Analysis Reveals Dynamic Changes of Whole Gut Microbiota in the Acute Phase of Intensive Care Unit Patients. Dig Dis Sci. 2016 Jun;61(6):1628-34. doi: 10.1007/s10620-015-4011-3. Epub 2015 Dec 29. PMID 26715502
- [Background] Kim D, Zeng MY, Nunez G. The interplay between host immune cells and gut microbiota in chronic inflammatory diseases. Exp Mol Med. 2017 May 26;49(5):e339. doi: 10.1038/emm.2017.24. PMID 28546562
- [Background] Czesnikiewicz-Guzik M, Muller DN. Scientists on the Spot: Salt, the microbiome, and cardiovascular diseases. Cardiovasc Res. 2018 Aug 1;114(10):e72-e73. doi: 10.1093/cvr/cvy171. No abstract available. PMID 30052920
- [Derived] Ding W, Zhang H, Wen J, Xiong G, Cheng M, Liu J, Zhao Y, Miao Q, Deng H, Xu Z, Mi L, Tan Z, Su L, Long Y, Ning K. A multi-omics analysis reveals a gut microbiome-LPC metabolic axis driving postoperative inflammation in cardiopulmonary bypass patients. Shock. 2025 Sep 18. doi: 10.1097/SHK.0000000000002722. Online ahead of print. PMID 41166145
- [Derived] Ding W, Liu J, Zhou X, Miao Q, Zheng H, Zhou B, Dou G, Tong Y, Long Y, Su L. Clinical Multi-Omics Study on the Gut Microbiota in Critically Ill Patients After Cardiovascular Surgery Combined With Cardiopulmonary Bypass With or Without Sepsis (MUL-GM-CSCPB Study): A Prospective Study Protocol. Front Med (Lausanne). 2020 Jul 8;7:269. doi: 10.3389/fmed.2020.00269. eCollection 2020. PMID 32733902